CLINICAL TRIAL: NCT00717379
Title: Open-Label, Randomized, Multicenter, Parallel-Group Efficacy and Safety Study of Tacrolimus Immunosuppressive Therapy After Kidney Transplantation
Brief Title: Study of Tacrolimus Immunosuppressive Therapy After Kidney Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Disclosure Office Europe, Astellas Pharma Europe BV
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRG-EC-2R01
Record Dates: First submitted 2008-07-16; First posted 2008-07-17 (Estimated); Last update posted 2009-04-15 (Estimated); Status verified 2009-04

CONDITIONS: Kidney Transplantation; Kidney Failure, Chronic; Renal Insufficiency, Chronic
Keywords: Organ Transplantation; Tacrolimus; Prograf; Kidney; Immunosuppression
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — Tacrolimus; Mycophenolic Acid; Methylprednisolone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): steroid regimen 1
  Interventions: Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Drug: Methylprednisolone or equivalent; Drug: Prednisone
- 2 (Experimental): steroid regimen 2
  Interventions: Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Drug: Methylprednisolone or equivalent; Drug: Prednisone

INTERVENTIONS:
Drug: Tacrolimus — oral
  Other Names: Prograf; FK506
Drug: Mycophenolate Mofetil — oral
  Other Names: MMF
Drug: Methylprednisolone or equivalent — oral
Drug: Prednisone — oral

SUMMARY:
To compare the efficacy and safety of Tacrolimus in combination with MMF and Steroids in two regimens of steroid in an adult kidney transplanted population.

ELIGIBILITY:
Inclusion Criteria:

* Female subject of childbearing potential must have a negative serum pregnancy test at enrolment and must agree to maintain effective birth control during the study
* Has an end stage kidney disease and is a suitable candidate for primary renal transplantation or retransplantation
* Subject is receiving a kidney transplant, from a cadaveric or living donor between 5 and 65 years of age with compatible AB0 blood type

Exclusion Criteria:

* Pregnant woman or breast-feeding mother
* Has an immunological high risk, defined as having a most recently measured PRA grade of > 50% within the previous six months
* Known allergy to the study drug or any of its components
* Requires ongoing dosing with a systemic immunosuppressive drug at study entry for any reason other than kidney transplantation
* Requires initial sequential or parallel therapy with immunosuppressive antibody preparation(s)
* Subject or donor is known to be HIV positive
* Has significant liver disease, defined as having during the past 28 days continuously elevated ASAT (SGOT) and/or ALAT (SGPT) levels greater than 3 times the upper value of the normal range of the investigational site
* Diagnosis of malignancy or history of malignancy, except non metastatic basal or squamous cell carcinoma of the skin that has been treated successfully
* Has significant, uncontrolled concomitant infections and/or severe diarrhoea, vomiting, or active peptic ulcer
* Previously received or is receiving an organ transplant other than kidney
* Receiving a graft from a non-heart-beating donor
* Cold ischemia time of the donor kidney >30 hours
* Any form of substance abuse, psychiatric disorder or condition which, in the opinion of the investigator, may complicate communication with the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Incidence and time to first biopsy-proven acute rejection | 6 months

SECONDARY OUTCOMES:
Overall frequency of acute rejection episodes within 6 months post transplantation | 6 months
Severity of biopsy proven acute rejections (BANFF criteria) within 6 months post transplantation | 6 months
Incidence of and time to first corticosteroid-resistant acute rejection | 6 months
Subject and graft survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — ZAO Astellas Pharma Russia
Locations (4):
- Russia (4):
  - Moscow
  - Omsk
  - Saint Petersburg
  - Volzskii